CLINICAL TRIAL: NCT02292303
Title: Randomized, Monocentric, Double-blind, 3-way-cross-over Clinical Trial to Determine the Bioavailability of Three Different Zinc Preparations
Brief Title: Clinical Trial to Determine the Bioavailability of Three Different Zinc Preparations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lesaffre International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTS812/14
Record Dates: First submitted 2014-11-07; First posted 2014-11-17 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2014-11

CONDITIONS: Zinc Deficiency
Keywords: Zinc/pharmacokinetics
MeSH Terms: interventions — Zinc Oxide; gluconic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- zinc-enriched yeast (Experimental): zinc-enriched yeast capsules
  Interventions: Dietary Supplement: zinc-enriched yeast
- zinc oxide (Active Comparator): zinc oxide capsules
  Interventions: Dietary Supplement: Zinc references
- zinc gluconate (Active Comparator): zinc gluconate capsules
  Interventions: Dietary Supplement: Zinc references

INTERVENTIONS:
Dietary Supplement: zinc-enriched yeast
  Arms: zinc-enriched yeast
Dietary Supplement: Zinc references
  Other Names: zinc oxide; zinc gluconate
  Arms: zinc gluconate; zinc oxide

SUMMARY:
The main objective of this clinical is to get information on pharmacokinetics of zinc-enriched yeast.The bioavailability of the yeast enriched with zinc will be compared to two selected zinc salts used in food supplements that are zinc oxide and zinc gluconate.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations
* Sex: female (premenopausal), male
* Age: 20 - 50 years
* BMI ≥19 or ≤30 kg/m²
* Non-smoker
* Subject is in good physical and mental health as established by medical history, physical examination, electrocardiogram, vital signs, results of biochemistry, hematology

Exclusion Criteria:

* Relevant history or presence of any medical disorder, potentially interfering with this trial
* For this trial clinically relevant abnormal laboratory, ECG, vital signs or physical findings at screening
* Migraine or regular headache, intense premenstrual symptoms
* Coffee consumption >3 cups / day
* Blood donation within 2 months prior to trial start or during trial
* Regular intake of mineral supplements within 4 weeks prior to trial start or during trial
* Chronic intake of substances affecting the intestinal absorption of zinc
* Vegetarians / vegans
* Drug-, alcohol- and medication abuses
* Known HIV-infection
* Known acute or chronic hepatitis B and C infection
* Relevant allergy or known hypersensitivity against compounds of the study preparations, for example lactose intolerance
* Known pregnancy, breast feeding or intention to become pregnant during the study
* Participation in another clinical trial within the last 4 weeks and concurrent participation in another clinical trial
* Not anticipating any planned changes in lifestyle for the duration of the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Comparison of pharmacokinetics parameters (AUC, Cmax and Tmax) between zinc-enriched yeast and zinc oxide. | Baseline (0 min); 30; 60; 90;120; 150; 180; 210; 240; 300 and 360 min

SECONDARY OUTCOMES:
Comparison of pharmacokinetics parameters (AUC, Cmax and Tmax) between zinc-enriched yeast and zinc gluconate. | Baseline (0 min); 30; 60; 90;120; 150; 180; 210; 240; 300 and 360 min